CLINICAL TRIAL: NCT00052910
Title: Phase III Intergroup Trial of Adjuvant Chemoradiation After Resection of Gastric or Gastroesophageal Adenocarcinoma
Brief Title: Chemotherapy and Radiation Therapy After Surgery in Treating Patients With Stomach or Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-80101; U10CA031946 (NIH); CDR0000258787 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Epirubicin; Fluorouracil; Leucovorin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive leucovorin calcium IV and fluorouracil (5-FU) IV on days 1-5 of courses 1, 3, and 4. Courses repeat every 28 days. During course 2, patients undergo radiotherapy 5 days a week and receive 5-FU IV continuously for 5 to 6 weeks. Patients rest for 28-35 days between course 2 and 3.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Radiation: radiation therapy
- Arm II (Experimental): Patients receive epirubicin IV over 3-15 minutes and cisplatin IV over 1 hour on day 1 and 5-FU IV continuously on days 1-21 during course 1. Beginning 1 week later, patients undergo radiotherapy 5 days a week and 5-FU IV continuously for 5 weeks. Patients rest for 28-35 days before beginning course 2 of chemotherapy. Patients then receive epirubicin, cisplatin, and 5-FU as in course 1. Treatment repeats every 21 days for 2 courses.
  Interventions: Drug: cisplatin; Drug: epirubicin hydrochloride; Drug: fluorouracil; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
  Arms: Arm II
Drug: epirubicin hydrochloride — Given IV
  Arms: Arm II
Drug: fluorouracil — Given IV
Drug: leucovorin calcium — Given IV
  Arms: Arm I
Radiation: radiation therapy — Given 5 days a week for 5 weeks

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy after surgery may kill any remaining tumor cells following surgery. It is not yet known which chemotherapy and radiation therapy regimen is more effective in treating stomach or esophageal cancer.

PURPOSE: Randomized phase III trial to compare two different chemotherapy and radiation therapy regimens in treating patients who have undergone surgery for stomach or esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival in patients with resected gastric adenocarcinoma treated with epirubicin, cisplatin, and infusional fluorouracil (5-FU) vs 5-FU bolus and leucovorin calcium before and after 5-FU plus radiotherapy.
* Compare disease-free survival and local and distant recurrence rates in these patients treated with these regimens.
* Correlate the expression of putative prognostic markers (including TS, ERCC-1, MSI, E-cadherin, EGFR, p27, COX-2, and c-erbB-2) with overall survival of patients treated with these regimens.
* Correlate specific germline polymorphisms related to chemotherapy metabolism and resistance (including UGT2B7 [epirubicin], GST [cisplatin], ERCCI [cisplatin], XRCC1 [cisplatin], TS [5-FU], DPD [5-FU], and EGFR polymorphisms) with treatment-related toxicity and overall survival of these patients.
* Correlate serum levels of insulin-like growth factor-1 (IGF-1), IGF-2, and IGF-binding protein 3 with overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to depth of tumor penetration (T1 or T2 vs T3 vs T4), lymph node involvement (0 vs 1-3), and extent of lymphadenectomy (D1 or D2 vs D0 or unknown). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive leucovorin calcium IV and fluorouracil (5-FU) IV on days 1-5 of courses 1, 3, and 4. Courses repeat every 28 days. During course 2, patients undergo radiotherapy 5 days a week and receive 5-FU IV continuously for 5 weeks. Patients rest for 28-35 days between course 2 and 3.
* Arm II: Patients receive epirubicin IV over 3-15 minutes and cisplatin IV over 1 hour on day 1 and 5-FU IV continuously on days 1-21 during course 1. Beginning 1 week later, patients undergo radiotherapy 5 days a week and receive 5-FU IV continuously for 5 weeks. Patients rest for 28-35 days before beginning course 2 of chemotherapy. Patients then receive epirubicin, cisplatin, and 5-FU as in course 1. Treatment repeats every 21 days for 2 courses.

Patients are followed every 3 months for 2 years, every 4 months for 2 years, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 824 patients will be accrued for this study.

ELIGIBILITY:
1. Required Tumor Parameters

   1.1 Patients must have histologically diagnosed adenocarcinoma of the stomach or gastroesophageal junction. Adenocarcinomas of the esophagus that are not involving the gastroesophageal junction are not eligible.

   1.2 Patients must have had en bloc resection of all known tumor. The surgical resection must have been done with a curative intent.

   1.3 Patients must have tumor extension beyond muscularis propria and/or nodal involvement without evidence of M1 disease.
   * Patients can have stages IB if there is evidence of either node-positive (N1) disease or tumor extension beyond the muscularis propria (i.e., T1, N1, M0 patients are eligible but patients with T2, N0, M0 are allowed only if there is extension beyond the muscularis propria).
   * Patients can have stages II, IIIA, IIIB or stage IV with M0 (i.e., T4N2M0).
   * Stages 0, IA, or any stage with M1 are not allowed. (see Appendix I for TNM staging guide).

   1.4 Patients with known unresected cancer, recurrent cancer, microscopic evidence of tumor at the distal or proximal line of stomach resection, noncontiguous resection of tumor, or M1 (metastatic) disease are ineligible.
2. Prior Therapy

   2.1 No prior therapy (except hormonal or biologic) for other malignancies is allowed except for adequately treated basal cell or squamous cell skin cancer, noninvasive carcinoma in situ which has been fully resected, or other cancer for which the patient has been disease free for five years.

   2.2 Patients who have had any previous chemotherapy or radiotherapy are ineligible.
3. Patient Characteristics

   3.1 Patients must have an ECOG (CTC) performance status of 0, 1 or 2.

   3.2 Patients are required to have an adequate total caloric intake to allow them to maintain their post-surgical body weight. Patients must have documentation of stable weight (or less than 2 pounds weight loss) for at least one week prior to registration.

   3.3 All patients must be evaluated by a radiation oncologist (prior to enrollment) to ensure that the patient is an appropriate candidate for radiation therapy.

   3.4 Patients may not have unilateral renal function (only one functioning kidney) as determined by CT scan with contrast, urogram, renal scan, or other study.

   3.5 Pregnant or lactating women may not participate. Men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method or practice abstinence while in this study.
   * The effects of therapeutic radiotherapy are known to be teratogenic.
   * The effects of Epirubicin, Cisplatin, and 5-FU on a developing human fetus at the recommended therapeutic dose are less well known.
   * For this reason and because DNA alkylating agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.
   * Should a woman become pregnant or suspect she is pregnant while participating on this study, she should inform her treating physician immediately. Because the risk of toxicity in nursing infants secondary to Epirubicin, Cisplatin, and 5-FU treatment of the mother is unknown but may be harmful, breastfeeding should be discontinued.

   3.6 Patients with any of the following cardiac conditions are ineligible:
   * Uncontrolled high blood pressure
   * Unstable angina
   * Symptomatic congestive heart failure
   * Myocardial infarction < 6 months prior to registration
   * Serious uncontrolled cardiac arrhythmia
   * New York Heart Association classification III or IV.

   3.7 No uncontrolled serious medical or psychiatric illness which would prevent compliance with treatment or adequate informed consent.

   3.8 Patients with active infectious process are ineligible.

   3.9 Patients with grade 2 or greater peripheral neuropathy at baseline are ineligible.
4. Required Initial Laboratory Values:

   * Granulocytes ≥ 1,500/μl
   * Platelet count ≥ 100,000/μl
   * Creatinine ≤ 1.5 mg/dl
   * Bilirubin ≤ 2.0 mg/dl
   * AST ≤ 3x upper limits of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2002-12; Primary Completion 2012-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Fuchs, MD, MPH, Study Chair — Dana-Farber Cancer Institute
Locations (535):
- United States (527):
  - Regional Medical Center, Anniston, Alabama
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Ben E. Owens Cancer Treatment Center at St. Bernard's Medical Center, Jonesboro, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Valley Medical Oncology, Fremont, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Community Hospital of the Monterey Peninsula Comprehensive Cancer Center, Monterey, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - San Francisco General Hospital Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Center for Cancer Care and Research at Watson Clinic, LLP, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Hematology Oncology Associates of Illinois - Berwyn, Berwyn, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Medical Consultants, PC at Ball Memorial Cancer Center, Muncie, Indiana
  - Community Hospital, Munster, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, PC - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Associates in Oncology and Hematology, Kensington, Maryland
  - Associates in Oncology and Hematology - Medical Center Drive, Rockville, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Morton Hospital & Medical Center, Taunton, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic, PA at Forrest General, Hattiesburg, Mississippi
  - Hematology & Oncology Clinic, Hattiesburg, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Christian Hospital Northeast Cancer Care Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - John F. Kennedy Medical Center, Edison, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - UPMC Cancer Center at Beaver Medical Center, Beaver, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Cancer Center at Jefferson Regional Medical Center, Clairton, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, PC at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Cancer Center at the John P. Murtha Pavilion, Johnstown, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - UPMC - Moon, Moon Township, Pennsylvania
  - UPMC Cancer Center - Natrona Heights, Natrona Heights, Pennsylvania
  - Jameson Memorial Hospital - North Campus, New Castle, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC St. Margaret, Pittsburgh, Pennsylvania
  - Mercy Cancer Institute at Mercy Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Passavant, Pittsburgh, Pennsylvania
  - St. Clair Memorial Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Washington Hospital Cancer Center, Washington, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island, Cranston, Rhode Island
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - AnMed Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Blue Ridge Medical Specialists, PC, Bristol, Tennessee
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Canada (8):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Result] Fuchs C, Tepper JE, Niedwiecki D, et al.: Postoperative adjuvant chemoradiation for gastric or gastroesophageal adenocarcinoma using epirubicin, cisplatin, and infusional (CI) 5-FU (ECF) before and after CI 5-FU and radiotherapy (RT): interim toxicity results from Intergroup trial CALGB 80101. [Abstract] American Society of Clinical Oncology 2006 Gastrointestinal Cancers Symposium, 26-28 January 2006, San Francisco, California. A-61, 2006.
- [Derived] Patel JN, Jiang C, Owzar K, Mulkey F, Luzum JA, Mamon HJ, Haller DG, Dragovich T, Alberts SR, Bjarnason G, Willet CG, Niedzwiecki D, Enzinger P, Ratain MJ, Fuchs C, McLeod HL. Pharmacogenetic study in gastric cancer patients treated with adjuvant fluorouracil/leucovorin or epirubicin/cisplatin/fluorouracil before and after chemoradiation on CALGB 80101 (Alliance). Pharmacogenet Genomics. 2021 Dec 1;31(9):215-220. doi: 10.1097/FPC.0000000000000442. PMID 34149004
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (5-FU/LV): Patients receive leucovorin calcium (LV) IV (20 mg/m^2 per day) and fluorouracil (5-FU) IV (425 mg/m^2 per day) on days 1-5 of courses 1, 3, and 4. Courses repeat every 28 days. During course 2, patients undergo radiotherapy 5 days a week and receive 5-FU IV continuously for 5 to 6 weeks. Patients rest for 28-35 days between course 2 and 3.
- Arm II (ECF): Patients receive epirubicin IV (50 mg/m^2) over 3-15 minutes and cisplatin IV (60 mg/m^2) over 1 hour on day 1 and 5-FU IV (200 mg/m^2 per day) continuously on days 1-21 during course 1. Beginning 1 week later, patients undergo radiotherapy 5 days a week and 5-FU IV continuously for 5 weeks. Patients rest for 28-35 days before beginning course 2 of chemotherapy. Patients then receive epirubicin, cisplatin, and 5-FU as in course 1. Treatment repeats every 21 days for 2 courses.
Period: Overall Study
Arm/Group | Arm I (5-FU/LV) | Arm II (ECF)
Started | 280 | 266
Completed | 280 | 266
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (5-FU/LV) | Arm II (ECF) | Total
Number analyzed (Participants) | 280 | 266 | 546
Age, Continuous [Median (Full Range); unit: years] | 59 [23 to 81] | 58 [29 to 83] | 58.6 [23 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 88 | 175
  Male | 193 | 178 | 371
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 17 | 38
  United States | 259 | 249 | 508

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from study enrollment to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From study enrollment until death from any cause; up to 3 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I (5-FU/LV) | Arm II (ECF)
Number analyzed (Participants) | 280 | 266
years | 3.6 [2.8 to 4.9] | 3.5 [2.5 to 5.0]
Statistical Analysis 1: Comparison: Arm I (5-FU/LV) vs Arm II (ECF); Test type: Superiority or Other; Cox Proportional Hazard = 0.99, 95% CI 2-sided [0.79 to 1.24] — Adjusted Hazard Ratio, ECF vs 5-FU/LV

2. Secondary Outcome: Disease Free Survival
Description: Disease free survival is defined as the time from the date of study enrollment to death or documented second primary tumor, or cancer recurrence.The distribution of disease free survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From the date of study enrollment until death or documented second primary tumor, or cancer recurrence; up to 4 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I (5-FU/LV) | Arm II (ECF)
Number analyzed (Participants) | 280 | 266
years | 2.7 [1.9 to 3.8] | 2.3 [1.5 to 3.1]
Statistical Analysis 1: Comparison: Arm I (5-FU/LV) vs Arm II (ECF); Test type: Superiority or Other; Cox Proportional Hazard = 1.03, 95% CI 2-sided [0.83 to 1.28] — Adjusted Hazard Ratio, ECF vs 5-FU/LV

ADVERSE EVENTS:
Arm/Group | Arm I (5-FU/LV) | Arm II (ECF)
All-Cause Mortality (participants affected / at risk) | 11/272 | 5/251
Serious Adverse Events (participants affected / at risk) | 62/272 | 42/251
Other Adverse Events (participants affected / at risk) | 258/272 | 234/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (5-FU/LV) (N=272) | Arm II (ECF) (N=251)
Blood disorder (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (7) | 8 (10)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Transfusion: Platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 2 (2) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 2 (2) | 0 (0)
Edema (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 27 (29) | 9 (9)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 31 (32) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 1 (1)
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 5 (5) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 5 (5) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 26 (27) | 5 (6)
Nausea (Gastrointestinal disorders) | 40 (41) | 19 (20)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (24) | 15 (16)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 1 (1)
Esophagus- Late RT Morbidity Scoring (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 32 (35) | 25 (28)
Fever (General disorders) | 2 (2) | 2 (3)
Heart- Late RT Morbidity Scoring (General disorders) | 1 (1) | 0 (0)
Joint- Late RT Morbidity Scoring (General disorders) | 0 (0) | 1 (1)
Lung-Late RT Morbidity Scoring (General disorders) | 0 (0) | 1 (1)
Mucous membrane-Late RT Morbidity Scoring (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2) | 4 (4)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 3 (3) | 1 (1)
Infection without neutropenia (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1)
Creatinine increased (Investigations) | 7 (7) | 3 (3)
INR increased (Investigations) | 2 (2) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 1 (1)
Leukocyte count decreased (Investigations) | 24 (25) | 19 (21)
Lymphocyte count decreased (Investigations) | 5 (5) | 4 (5)
Neutrophil count decreased (Investigations) | 25 (26) | 20 (22)
Platelet count decreased (Investigations) | 14 (15) | 9 (10)
Serum cholesterol increased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 6 (6) | 7 (7)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 27 (29) | 16 (18)
Blood glucose increased (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 16 (16) | 9 (10)
Serum albumin decreased (Metabolism and nutrition disorders) | 6 (6) | 2 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 11 (12) | 3 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6) | 4 (4)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 7 (8) | 4 (4)
Thrombosis (Vascular disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (5-FU/LV) (N=272) | Arm II (ECF) (N=251)
Blood disorder (Blood and lymphatic system disorders) | 2 (4) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (11) | 8 (10)
Hemoglobin decreased (Blood and lymphatic system disorders) | 80 (165) | 81 (180)
Hemoglobin for leukemia studies (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 6 (6)
Cardiac pain (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Edema (Cardiac disorders) | 5 (5) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (4) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Hearing test abnormal (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 3 (6) | 2 (3)
Flashing vision (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (3) | 1 (1)
Watering eyes (Eye disorders) | 2 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 109 (186) | 94 (141)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 4 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 37 (54) | 40 (59)
Diarrhea (Gastrointestinal disorders) | 162 (313) | 120 (227)
Dry mouth (Gastrointestinal disorders) | 4 (6) | 5 (6)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 18 (24) | 21 (35)
Dysphagia (Gastrointestinal disorders) | 24 (29) | 23 (37)
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 11 (14) | 13 (15)
Fistula of small intestine (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 10 (13) | 4 (9)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 7 (8) | 7 (9)
Gastrointestinal disorder (Gastrointestinal disorders) | 8 (9) | 7 (8)
Hemorrhoids (Gastrointestinal disorders) | 1 (3) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 2 (2)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis due to radiation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 155 (248) | 107 (168)
Nausea (Gastrointestinal disorders) | 192 (390) | 176 (425)
Oral pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (4)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 123 (191) | 120 (209)
Bladder- Late RT Morbidity Scoring (General disorders) | 0 (0) | 3 (3)
Bone - Late RT Morbidity Scoring (General disorders) | 0 (0) | 2 (2)
Brain- Late RT Morbidity Scoring (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 5 (7) | 8 (10)
Chills (General disorders) | 3 (5) | 3 (4)
Edema limbs (General disorders) | 3 (3) | 7 (10)
Esophagus- Late RT Morbidity Scoring (General disorders) | 19 (63) | 19 (32)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 201 (493) | 190 (503)
Fever (General disorders) | 10 (11) | 6 (6)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
General symptom (General disorders) | 2 (2) | 3 (4)
Heart- Late RT Morbidity Scoring (General disorders) | 3 (4) | 4 (7)
Ill-defined disorder (General disorders) | 2 (2) | 1 (1)
Joint- Late RT Morbidity Scoring (General disorders) | 2 (2) | 1 (1)
Kidney-Late RT Morbidity Scoring (General disorders) | 3 (3) | 3 (6)
Larynx-Late RT Morbidity Scoring (General disorders) | 2 (2) | 1 (2)
Liver-Late RT Morbidity Scoring (General disorders) | 6 (17) | 4 (7)
Localized edema (General disorders) | 1 (1) | 1 (1)
Lung-Late RT Morbidity Scoring (General disorders) | 8 (11) | 6 (14)
Mucous membrane-Late RT Morbidity Scoring (General disorders) | 3 (3) | 4 (5)
Pain (General disorders) | 19 (31) | 23 (32)
Pericardial pain (General disorders) | 0 (0) | 1 (1)
Radiation-Other(Specify,_____) (General disorders) | 17 (24) | 11 (28)
Salivary glands-Late RT Morbidity Scoring (General disorders) | 1 (1) | 1 (1)
Skin-Late RT Morbidity Scoring (General disorders) | 6 (6) | 3 (3)
Small/Large intestine-Late RT Morbidity Scoring (General disorders) | 12 (16) | 12 (23)
Subcutaneous tissue-Late RT Morbidity Scoring (General disorders) | 1 (1) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 3 (6) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 2 (2) | 0 (0)
Bladder infection (Infections and infestations) | 2 (4) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (2) | 5 (6)
Device related infection (Infections and infestations) | 1 (2) | 2 (2)
Esophageal infection (Infections and infestations) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 10 (13) | 1 (1)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 4 (4) | 2 (3)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 6 (6) | 7 (7)
Infectious colitis (Infections and infestations) | 3 (3) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 2 (3)
Paranasal sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 2 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 2 (3)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 2 (2) | 2 (3)
Wound-infectious (Infections and infestations) | 2 (2) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 23 (26) | 16 (21)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative gastrointestinal injury - Appendix (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 4 (4) | 1 (1)
Alanine aminotransferase increased (Investigations) | 21 (34) | 22 (36)
Alkaline phosphatase (Investigations) | 4 (8) | 5 (7)
Alkaline phosphatase increased (Investigations) | 22 (32) | 17 (23)
Amylase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 36 (54) | 28 (36)
Blood bilirubin increased (Investigations) | 16 (22) | 7 (8)
Coagulopathy (Investigations) | 5 (6) | 0 (0)
Creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 22 (29) | 17 (34)
Gamma-glutamyltransferase increased (Investigations) | 2 (4) | 2 (4)
Haptoglobin decreased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 4 (5) | 2 (2)
Laboratory test abnormal (Investigations) | 3 (5) | 4 (4)
Leukocyte count decreased (Investigations) | 177 (409) | 177 (458)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 39 (75) | 32 (67)
Neutrophil count decreased (Investigations) | 178 (333) | 166 (361)
Platelet count decreased (Investigations) | 92 (167) | 74 (145)
Weight gain (Investigations) | 0 (0) | 3 (3)
Weight loss (Investigations) | 59 (96) | 51 (90)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 148 (279) | 140 (294)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 41 (66) | 47 (77)
Dehydration (Metabolism and nutrition disorders) | 33 (45) | 31 (45)
Serum albumin decreased (Metabolism and nutrition disorders) | 32 (40) | 28 (44)
Serum calcium decreased (Metabolism and nutrition disorders) | 28 (38) | 23 (28)
Serum glucose decreased (Metabolism and nutrition disorders) | 5 (8) | 10 (13)
Serum magnesium decreased (Metabolism and nutrition disorders) | 5 (7) | 10 (17)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 31 (44) | 26 (43)
Serum potassium increased (Metabolism and nutrition disorders) | 7 (8) | 4 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 24 (32) | 14 (24)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (14) | 6 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (12) | 11 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (7)
Ataxia (Nervous system disorders) | 2 (2) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 15 (18) | 22 (33)
Dysgeusia (Nervous system disorders) | 27 (41) | 20 (39)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 13 (17) | 17 (23)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (4)
Neurological disorder NOS (Nervous system disorders) | 2 (4) | 0 (0)
Neuropathy - cranial (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 34 (55) | 38 (62)
Syncope (Nervous system disorders) | 3 (3) | 4 (4)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 2 (3) | 3 (4)
Anxiety (Psychiatric disorders) | 5 (7) | 12 (27)
Depression (Psychiatric disorders) | 9 (13) | 18 (29)
Euphoria (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 17 (22) | 16 (23)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (1) | 1 (2)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 4 (5)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (3)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 2 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (35) | 18 (25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 7 (12)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 7 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (37) | 49 (104)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Dermatology (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (12) | 6 (8)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 36 (52) | 46 (75)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 14 (21)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (11) | 4 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 30 (39) | 13 (16)
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 7 (10) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 (8) | 7 (9)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (7)
Flushing (Vascular disorders) | 4 (7) | 2 (3)
Hemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Vascular disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 4 (5)
Hypotension (Vascular disorders) | 7 (10) | 11 (14)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 6 (7) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes